CLINICAL TRIAL: NCT03796910
Title: A Two-part, Randomized, Double-blind, Placebo-controlled, First-In-Human, Phase I Study of the Safety, Tolerability, and Pharmacokinetics of SPR720 Following Administration of Single and Multiple Ascending Oral Doses in Healthy Volunteers
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of SPR720 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR720-101
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: safety; tolerability; pharmacokinetics; SPR720
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, single and multiple ascending dose (SAD and MAD) trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized in a 3:1 ratio to receive SPR720 or placebo. The randomization code will produced by Simbec using the PROC PLAN procedure of SAS® version 9.3 or higher. The randomization code will include 2 dose-leaders (1 active:1 placebo) in each cohort who will be randomized prior to the remainder of the cohort. The allocation to SPR720 or placebo will be performed using a block randomization algorithm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SPR720 for SAD (Experimental): 6 out of 8 subjects per cohort will be randomized to receive SPR720
  Interventions: Drug: SPR720 for SAD
- Placebo for SAD (Placebo Comparator): 2 out of 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo for SAD
- SPR720 for MAD (Experimental): 6 out of 8 subjects per cohort will be randomized to receive SPR720
  Interventions: Drug: SPR720 for MAD
- Placebo for MAD (Placebo Comparator): 2 out of 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo for MAD

INTERVENTIONS:
Drug: SPR720 for SAD — Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 8 dose ascending cohorts) to receive either SPR720 or placebo. The study drug (SPR720 or placebo) will be administered as a single dose.
  Other Names: SPR720 Oral Capsule
  Arms: SPR720 for SAD
Drug: Placebo for SAD — Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 8 dose ascending cohorts) to receive either SPR720 or placebo. The study drug (SPR720 or placebo) will be administered orally as a single dose.
  Other Names: Placebo oral Capsule
  Arms: Placebo for SAD
Drug: SPR720 for MAD — Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 3 cohorts) to receive either SPR720 or placebo. The study drug (SPR720 or placebo) will be administered orally for a total of 7 (or 14) days of dosing.
  Other Names: SPR720 Oral Capsule
  Arms: SPR720 for MAD
Drug: Placebo for MAD — Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 3 cohorts) to receive either SPR720 or placebo. The study drug (SPR720 or placebo) will be administered orally for a total of 7 (or 14) days of dosing
  Other Names: Placebo Oral Capsule
  Arms: Placebo for MAD

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics (PK) following single and multiple ascending dose administration of SPR720 administered orally in healthy volunteers.

DETAILED DESCRIPTION:
This is a single-center, phase I, randomized, double-blind, placebo-controlled, first-in-man study. Up to 120 healthy volunteers may be enrolled in this 2-part, multi-cohort study. In both Part 1 and Part 2, sequential cohorts will be exposed to increasing doses of SPR720. Each cohort will enrol 8 subjects, randomized (3:1) to receive SPR720 (6 subjects) or placebo (2 subjects). Each subject will be assigned to only one cohort.

In Part 1 single ascending dose (SAD):

A single oral dose of SPR720 (n=6) or placebo (n=2) will be administered to 8 subjects at an initial dose level of 100 mg. Additional cohorts of 8 subjects will be enrolled to investigate increasing doses of SPR720 ranging from 250 mg to 3000 mg. All subjects will receive SPR720 (or placebo) by oral administration in the fasted state. One Part 1 cohort (the Food Effect Cohort) will receive an additional single dose of SPR720 (or placebo) in the fed state.

Part 2 multiple ascending dose (MAD):

SPR720 (or placebo) will be administered to approximately 3 planned dose cohorts of 8 subjects each. Subjects will receive SPR720 (or placebo) orally once daily for 7 (or 14) consecutive days starting with a planned initial dose of 500 mg. Additional cohorts of 8 subjects will be enrolled to investigate repeated daily doses of SPR720 ranging from 1000 mg to 1500 mg.

For both Part 1 and Part 2, a Safety Monitoring Group (SMG) will review cumulative safety and PK data from each cohort before proceeding to the next cohort/dose level. Doses to be evaluated in each subsequent cohort may be modified by the SMG based on review of safety and PK data from preceding cohorts. Part 2 will run concurrent with Part 1 and will be initiated following SMG review of safety and PK data for the corresponding Part 1 dose level cohort.

Part 1 will be conducted in up to 64 subjects (8 planned dose cohorts of 8 subjects each). Part 2 will be conducted in up to 24 subjects (3 planned dose cohorts of 8 subjects each); additional cohorts of 8 subjects each (up to 16 additional subjects) may be enrolled in either Part if further investigation of SPR720 is required.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

1. Healthy adult male or female of non-childbearing potential,18 to 55 or ≥ 65 years of age (inclusive) at the time of screening;
2. Body mass index (BMI) ≥ 18.5 and ≤ 32 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive). BMI = body weight (kg) / [height (m)]2 (subjects 18 to 55 years of age); Body mass index (BMI) ≥ 18 and ≤ 32 (kg/m2) and weight between 50.0 and 100.0 kg (inclusive). BMI = body weight (kg) / [height (m)]2 (subjects 65 years of age and older);
3. Medically healthy without clinically significant (CS) abnormalities as assessed by the Principal Investigator (or deputy) based on the following at screening assessments:

   a. Detailed medical history, complete physical examination, vital signs, 12-lead ECG, hematology, blood chemistry and urinalysis laboratory variables;
4. Willing and able to provide written informed consent;
5. Willing and able to comply with all study assessments and adhere to the protocol schedule;
6. If female, must be non-lactating and be of non-childbearing potential;
7. If male, must agree to not donate sperm for 90 days after the last dose of study drug and, if engaging in vaginal sexual intercourse with a female partner of childbearing potential, agree to use a condom with spermicide in addition to requesting the female partner use a highly effective method of birth control (e.g. intrauterine device, diaphragm with spermicide, hormonal contraceptives) throughout the duration of the study and for 90 days after the last dose of study drug. This criterion also applies to males who have had a vasectomy.

KEY EXCLUSION CRITERIA:

1. History or presence of any clinically significant disease state in any body system, as assessed by the Principal Investigator (or deputy), that may affect the outcome of the study or compromise the safety of the subject;
2. Subjects who do not have suitable veins for multiple venipunctures/cannulation as assessed by the Principal Investigator (or deputy) at screening;
3. Subjects who are unable to demonstrate the ability to swallow a "dummy" capsule (i.e., an empty gelatin capsule) of the size proposed for administration in a particular cohort/dose level;
4. History of any clinically significant acute illness or surgery within the previous three months;
5. History of chronic gastritis, gastrointestinal tract disorders, including Clostridium difficile infection; chronic liver or biliary disease;
6. History of seizure disorder, except for febrile seizures in childhood;
7. Documented history of significant hypersensitivity reaction or anaphylaxis to any medication;
8. History of significant allergic disease requiring treatment; allergic rhinitis (hay fever) is allowed unless it has required medication for treatment or prophylaxis within the 14 days prior to randomization;
9. Clinically significant screening ECG findings as assessed by the investigator;
10. Subject or family history of cardiac arrhythmia, prolonged QT syndrome, Torsades de pointes, unexplained sudden cardiac arrest or syncope, sick sinus syndrome or other clinically relevant cardiac disease;
11. Clinically significant abnormalities in vital signs at screening and/or prior to randomization;
12. Clinically significant screening laboratory abnormalities;
13. History or suspicion of routine or chronic drug or alcohol abuse or dependence within 1 year prior to randomization, and/or positive urine drug testing at screening or check-in (Day -1);
14. Reported consumption of alcoholic beverages > 21 units per week on average (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits); positive alcohol urine test at check in (Day -1);
15. Use of tobacco, nicotine, or nicotine replacement products within 30 days prior to randomization or planned use during the study; positive carbon monoxide breath test at check in (Day -1);
16. Use of any prescription or non-prescription medication, including herbal products, vitamins and vaccines within 7 days (or 5 half-lives whichever is longer) prior to randomization or planned use during the study period;
17. Consumption of grapefruit or grapefruit-containing products in the 7 days prior to randomization;
18. Donation of more than 500 mL of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events assessments after single and multiple dose administration at baseline and repeatedly until study completion [Safety and Tolerability] | Day 1 through last follow-up visit (5-7 days after last dose)
  Incidence and severity of AEs

SECONDARY OUTCOMES:
Assessment of Pharmacokinetic Parameter (plasma): Cmax measurement | From Day 1 pre-dose to 48 hours post last dose
  Maximum concentration of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): CmaxSS measurement | From Day 1 pre-dose to 48 hours post last dose
  Maximum concentration of study drug in plasma at steady state
Assessment of Pharmacokinetic Parameter (plasma): CminSS | From Day 1 pre-dose to 48 hours post last dose
  Lowest concentration of study drug in a dosing interval in plasma
Assessment of Pharmacokinetic Parameter (plasma): Ctrough | From Day 1 pre-dose to 48 hours post last dose
  Concentration of study drug at the end of the dosing interval in plasma
Assessment of Pharmacokinetic Parameter (plasma): CavSS | From Day 1 pre-dose to 48 hours post last dose
  Average concentration of study drug in plasma during a dosing interval
Assessment of Pharmacokinetic Parameter (plasma): Tmax | From Day 1 pre-dose to 48 hours post last dose
  The time to maximum observed concentration of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): kel | From Day 1 pre-dose to 48 hours post last dose
  Elimination rate constant of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): t1/2 | From Day 1 pre-dose to 48 hours post last dose
  Terminal elimination half-life of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): AUC0-24 | From Day 1 pre-dose to 48 hours post last dose
  Area under the concentration-time curve (AUC) of study drug in plasma from 0 to 24 hours post dose (dose escalation)
Assessment of Pharmacokinetic Parameter (plasma): AUC0-tau | From Day 1 pre-dose to 48 hours post last dose
  Area under the concentration-time curve (AUC) from 0 to tau, where tau is the dosing interval (multiple dose only) of study drug in plasma
Assessment of Parameter (plasma): AUC0-t | From Day 1 pre-dose to 48 hours post last dose
  Area under the concentration-time curve (AUC) of study drug in plasma from the time of dosing to the time of the last measurable concentration
Assessment of Pharmacokinetic Parameter (plasma): AUC0-inf | From Day 1 pre-dose to 48 hours post last dose
  AUC extrapolated to infinity of study drug in plasma
Assessment of Parameter (plasma): AUC%extrapolated | From Day 1 pre-dose to 48 hours post last dose
  Residual area of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): Degree of fluctuation | From Day 1 pre-dose to 48 hours post last dose
  (Cmax-Cmin)/Cavss of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): Swing | From Day 1 pre-dose to 48 hours post last dose
  (Cmaxss-Cminss)/Cminss of study drug in plasma
Assessment of Pharmacokinetic Parameter (urine): SPR719 | From Day 1 pre-dose to 24 hours post last dose
  amount of SPR719 excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Ltd., Merthyr Tydfil, Mid Glamorgan, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talley AK, Thurston A, Moore G, Gupta VK, Satterfield M, Manyak E, Stokes S, Dane A, Melnick D. First-in-Human Evaluation of the Safety, Tolerability, and Pharmacokinetics of SPR720, a Novel Oral Bacterial DNA Gyrase (GyrB) Inhibitor for Mycobacterial Infections. Antimicrob Agents Chemother. 2021 Oct 18;65(11):e0120821. doi: 10.1128/AAC.01208-21. Epub 2021 Sep 7. PMID 34491803